CLINICAL TRIAL: NCT04322292
Title: A Phase Ⅰ Study Evaluating Safety and Efficacy of C-CAR088 Treatment in Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of BCMA-directed CAR-T Cells Treatment in Subjects With r/r Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QT2019007
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2024-05

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- C-CAR088 (Experimental): Lymphocytes will be transduced with lentiviral vector containing CAR-BCMA gene.
  Interventions: Drug: C-CAR088

INTERVENTIONS:
Drug: C-CAR088 — Autologous BCMA-directed CAR-T cells, single infusion intravenously at a target dose of 1.0-9.0 x 10^6 anti-BCMA CAR+T cells/kg.
  Other Name: CBM.BCMA Chimeric Antigen Receptor T cell.

SUMMARY:
This is a single-center, non-randomized and dose-escalation study to evaluate the safety and efficacy of C-CAR088 in relapsed or refractory multiple myeloma patient.

DETAILED DESCRIPTION:
The study will include the following sequential phases: Screening, Pre- Treatment (Cell Product Preparation, Lymphodepleting Chemotherapy), C-CAR088 infusion and Follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old, male or female;
2. The patient volunteered to participate in the study, and he or his legal guardian signed the Informed Consent;
3. Meet the internationally accepted Criteria for the diagnosis of multiple myeloma (IMWG diagnostic criteria 2014);
4. Patients with a clear diagnosis of relapsed or refractory multiple myeloma；
5. The patient have one or more measurable multiple myeloma lesion, must include one of the following conditions:

   * Serum M protein≥1.0 g/dL(10g/L)
   * Urine M protein≥200 mg/24h
   * Serum free light chain(sFLC): κ/λ FLC ratio is abnormal and affected FLC ≥10mg / dL
6. Bone marrow sample is confirmed as BCMA-positive by flow cytometry or pathological examination;
7. ECOG scores 0 - 1;
8. Echocardiography showed normal diastolic function, left ventricular ejection fraction (LVEF) ≥50%, and no severe arrhythmia;
9. No active pulmonary infections, normal pulmonary function and oxygen saturation ≥ 92% on room air.
10. Absolute neutrophil count ≥1.0 × 109 / L, platelet count ≥50 × 109 / L; total serum bilirubin ≤1.5mg / dl; serum ALT or AST less than 2.5 times the upper limit of normal; serum creatinine ≤2.0mg / dl;
11. No contraindications of peripheral blood apheresis;
12. Expected survival time > 12 weeks;.
13. Female subjects of childbearing age must have a negative urine / blood pregnancy test within 7 days before cell therapy and not be in lactation; female or male subjects of childbearing age need to take effective contraception throughout the study.

Exclusion Criteria:

1. Have a history of allergy to cellular products;
2. Presence of clinically significant cardiovascular disease;
3. A history of craniocerebral trauma, consciousness disorder, epilepsy, severe cerebral ischemia or hemorrhagic disease;
4. Need to use any anticoagulant (except aspirin);
5. Patients requiring urgent treatment due to tumor progression or spinal cord compression;
6. Patients with CNS metastasis or symptoms of CNS involvement;
7. After allogeneic hematopoietic stem cell transplantation;
8. Plasma cell leukemia;
9. Received systemic anti-tumor treatment within 2 weeks before apheresis, and within 1 week before apheresis, prednisone (or equivalent amount of other corticosteroids) was applied in excess of 5 mg/d ;
10. Patients with autoimmune diseases, immunodeficiency, or other immunosuppressive agents;
11. Uncontrolled active infection;
12. Have used any CAR T cell products or other genetically modified T cell therapy before;
13. Hepatitis B or hepatitis C virus infection (including carriers), syphilis, as well as acquired, congenital immune deficiency diseases, including but not limited to HIV infected persons;
14. Have a history of alcoholism, drug addiction and mental illness;
15. Participated in any other clinical trial within 1 months;
16. The investigators believe that there are other circumstances that are not suitable for the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2022-09-22 (Actual)

PRIMARY OUTCOMES:
Safety: The incidence of treatment-emergent adverse events (TEAEs) | 30 days
  The incidence of treatment-emergent adverse events (TEAEs)

SECONDARY OUTCOMES:
Overall response rate (ORR) | 12 months
  ORR(including sCR / CR / VGPR / PR, based on IMWG 2016 efficacy evaluation criteria)
Progression free survival (PFS) | 6 months、12 months
  PFS(based on IMWG 2016 efficacy evaluation criteria)
The CART cell duration in vivo | 12 months
  The copys of BCMA-CART DNA in peripheral blood with qPCR method
The soluble BCMA changes in peripheral blood | 12 months
  The amount of soluble BCMA in peripheral blood with ELISA method

CONTACTS AND LOCATIONS:
Locations (1):
- InstituteHBDH, Tianjin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qu X, An G, Sui W, Wang T, Zhang X, Yang J, Zhang Y, Zhang L, Zhu D, Huang J, Zhu S, Yao X, Li J, Zheng C, Zhu K, Wei Y, Lv X, Lan L, Yao Y, Zhou D, Lu P, Qiu L, Li J. Phase 1 study of C-CAR088, a novel humanized anti-BCMA CAR T-cell therapy in relapsed/refractory multiple myeloma. J Immunother Cancer. 2022 Sep;10(9):e005145. doi: 10.1136/jitc-2022-005145. PMID 36100310